CLINICAL TRIAL: NCT01510028
Title: A Phase I/II Multicenter Open-label Dose Escalation Study of HGT-1110 Administered Intrathecally in Children With Metachromatic Leukodystrophy
Brief Title: Multicenter Study of HGT-1110 Administered Intrathecally in Children With Metachromatic Leukodystrophy (MLD)
Acronym: IDEAMLD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HGT-MLD-070; 2011-002044-28 (EudraCT Number); U1111-1153-1422 (Other: WHO)
Record Dates: First submitted 2011-12-14; First posted 2012-01-13 (Estimated); Results first posted 2018-10-15 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Metachromatic Leukodystrophy (MLD)
Keywords: Intrathecal Drug Delivery Device (IDDD); Recombinant human arylsulfatase A (rhASA); Metachromatic Leukodystrophy (MLD)
MeSH Terms: conditions — Leukodystrophy, Metachromatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (10 mg) (Experimental): 6 patients treated with HGT-1110 10 mg EOW by IT injection
  Interventions: Biological: Recombinant human arylsulfatase A
- Cohort 2 (30 mg) (Experimental): 6 patients treated with HGT-1110 30 mg EOW by IT injection
  Interventions: Biological: Recombinant human arylsulfatase A
- Cohort 3 (100 mg) (Experimental): 6 patients treated with HGT-1110 100 mg EOW by IT injection
  Interventions: Biological: Recombinant human arylsulfatase A
- Cohort 4 (100 mg) (Experimental): 6 patients treated with HGT-1110 100 mg EOW by IT injection
  Interventions: Biological: Recombinant human arylsulfatase A

INTERVENTIONS:
Biological: Recombinant human arylsulfatase A — 6 patients treated with HGT-1110 EOW by IT injection
  Other Names: HGT-1110; rhASA

SUMMARY:
The purpose of this study is to determine the safety of ascending doses of HGT-1110 administered by intrathecal (IT) injection for 38 weeks (20 injections) in children with metachromatic leukodystrophy (MLD).

DETAILED DESCRIPTION:
Metachromatic leukodystrophy (MLD) is an inherited, autosomal recessive disorder of lipid metabolism characterized by deficient activity of the lysosomal enzyme, arylsulfatase A (ASA). MLD is a rare disease that occurs in most parts of the world. The estimated overall incidence of the disease in the western world is approximately 1 in 100,000 live births that varies by geographic location. There are no approved therapies for MLD.

This is a multicenter, open-label, dose-escalation study designed to evaluate the safety of up to 3 dose levels (10, 30, or 100 mg) of HGT-1110 administered via an intrathecal drug delivery device (IDDD) every other week (EOW) for a total of 38 weeks (20 injections, Weeks 0 to 38) to children with MLD. The study also includes the assessment of HGT-1110 drug product produced with a revised drug substance manufacturing process (referred to as Process B) in a fourth cohort (Cohort 4). Approximately 24 patients will be enrolled and will receive treatment of HGT-1110. Patients will be sequentially enrolled into 4 dose cohorts, approximately 6 patients each. Patient enrollment will be staggered in this study to facilitate adequate safety monitoring per dose cohort.

ELIGIBILITY:
Inclusion

For Cohorts 1-4:

1. Confirmed diagnosis of metachromatic leukodystrophy by both:

   * Arylsulfatase A (ASA) deficiency by assay in leukocytes AND
   * Elevated sulfatide in urine
2. Appearance of the first symptoms of disease at or before 30 months of age.

   For Cohorts 1-3 only:
3. Ambulatory at the time of screening. The minimum level of function required to meet this criterion is defined as the ability to walk forward 10 steps with one hand held.
4. The patient is less than 12 years of age at the time of screening.

   For Cohort 4 only:

   3.1 Minimum motor function requirements:
   1. A total GMFM-88 (percent) score ≥40 at the screening examination and a total GMFM-88 (percent) score ≥35 at the baseline examination, AND
   2. GMFM-88 Dimension E: Walking, Running & Jumping, item 68 ("walk forward 10 steps with one hand held") score of at least 1 "initiates" at the screening and baseline examinations (if applicable).

   4.1 The patient is less than 8 years of age at the time of screening.

   For Cohorts 1-4:
5. Neurological signs of MLD must be present at the screening examination.
6. The patient and his/her parent/representative(s) must have the ability to comply with the clinical protocol.
7. Patient's parent(s) or legally authorized representative(s) must provide written informed consent prior to performing any study-related activities. Study-related activities are any procedures that would not have been performed during normal management of the patient.

Exclusion Criteria:

Patients will be excluded from the study if there is evidence or history of any of the following criteria at screening:

For Cohorts 1-4:

1. History of hematopoietic stem cell transplantation (HSCT).
2. The patient has any known or suspected hypersensitivity to anesthesia or is thought to be at an unacceptably high risk for anesthesia due to airway compromise or other conditions.
3. Any other medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the trial.
4. The patient is enrolled in another clinical study that involves the use of any investigational product (drug or device) other than HGT-1110 or the IDDD used in this study within 30 days prior to study enrollment or at any time during the study.
5. The patient is pregnant or breastfeeding.
6. The patient has a condition that is contraindicated as described in the SOPH-A-PORT

Mini S IDDD Instructions for Use (IFU), including:

1. The patient has had, or may have, an allergic reaction to the materials of construction of the SOPH-A-PORT Mini S device.
2. The patient's body size is too small to support the size of the SOPH-A-PORT Mini S Access Port, as judged by the Investigator.
3. The patient has a known or suspected local or general infection.
4. The patient is at risk of abnormal bleeding due to a medical condition or therapy.
5. The patient has one or more spinal abnormalities that could complicate safe implantation or fixation.
6. The patient has a functioning CSF shunt device.
7. The patient has shown an intolerance to an implanted device.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2012-02-02 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2017-01-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- The Children's Hospital at Westmead, Westmead, Australia
- Rigshospitalet, Copenhagen, Denmark
- Hopital de Bicetre, Le Kremlin-Bicêtre, Île-de-France Region, France
- Center for Pediatric Clinical Studies, Tübingen, Baden-Wurttemberg, Germany
- Osaka University Hospital, Suita, Japan

IPD SHARING:
Plan to Share IPD: No
- De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites, …)

REFERENCES:
- [Derived] I Dali C, Sevin C, Krageloh-Mann I, Giugliani R, Sakai N, Wu J, Wasilewski M. Safety of intrathecal delivery of recombinant human arylsulfatase A in children with metachromatic leukodystrophy: Results from a phase 1/2 clinical trial. Mol Genet Metab. 2020 Sep-Oct;131(1-2):235-244. doi: 10.1016/j.ymgme.2020.07.002. Epub 2020 Jul 16. PMID 32792226

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 5 main sites for cohorts 1 to 3 in Brazil, Denmark, Germany, France, and Australia and 3 main sites for cohort 4 in Denmark, France, and Germany between 02 February 2012 (first participant first visit) and 20 January 2017 (last participant last visit).
Pre-assignment Details: A total of 34 participants were screened and 24 participants were enrolled in the study. Out of which 23 participants completed the study.
Groups:
- SHP611 10 mg (Process A): Participants received 10 milligram (mg) dose of SHP611 (HGT-1110, recombinant human arylsulfatase A [rhASA]) every other week (EOW) by intrathecal drug delivery device (IDDD) for 38 weeks. In this cohort, participants received SHP611 produced with the original drug substance manufacturing process referred to as Process A.
- SHP611 30 mg (Process A): Participants received 30 mg dose of SHP611 (HGT-1110, rhASA) EOW by IDDD for 38 weeks. In this cohort, participants received SHP611 produced with the original drug substance manufacturing process referred to as Process A.
- SHP611 100 mg (Process A): Participants received 100 mg dose of SHP611 (HGT-1110, rhASA) EOW by IDDD for 38 weeks. In this cohort, participants received SHP611 produced with the original drug substance manufacturing process referred to as Process A.
- SHP611 100 mg (Process B): Participants received 100 mg dose of SHP611 (HGT-1110, rhASA) EOW by IDDD for 38 weeks. In this cohort, participants received SHP611 produced with the revised drug substance manufacturing process referred to as Process B.
Period: Overall Study
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Started | 6 | 6 | 6 | 6
Completed | 5 | 6 | 6 | 6
Not Completed | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety set consisted of participants who received at least 1 dose of investigational product or underwent device implant surgery.
Groups:
- SHP611 10 mg (Process A): Participants received 10 mg dose of SHP611 (HGT-1110, rhASA) EOW by IDDD for 38 weeks. In this cohort, participants received SHP611 produced with the original drug substance manufacturing process referred to as Process A.
- Total: Total of all reporting groups
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 24
Age, Continuous [Mean (Standard Deviation); unit: Months] | 31.5 (11.50) | 47.3 (20.23) | 52.2 (31.17) | 48.5 (24.22) | 44.9 (22.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 1 | 2 | 9
  Male | 3 | 3 | 5 | 4 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 5 | 4 | 2 | 4 | 15
  Race: Asian | 0 | 0 | 4 | 0 | 4
  Race: Other | 1 | 2 | 0 | 2 | 5
  Ethnicity: Not Hispanic or Latino | 6 | 6 | 6 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) by Type and Severity
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were defined as all AEs that occurred at or after the first dose of the investigational product or device implant surgery (whichever occurred earlier) and through the last follow-up date. Drug-related and device-related types of TEAEs were analyzed and reported. The severity of AEs was assessed by the investigator using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.0 grading scale. Severity of all AEs or SAEs was recorded as grade 1, 2, 3, 4, or 5 corresponding, respectively, to a severity of mild, moderate, severe, life-threatening, or fatal. Here SDI refers to surgical device implantation.
Time Frame: From start of study treatment up to Week 42
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  TEAE | 6 | 6 | 6 | 6
  SHP611-related TEAE | 3 | 4 | 4 | 2
  SDI-related TEAE | 5 | 3 | 4 | 4
  IDDD-related TEAE | 3 | 3 | 4 | 0
  SOPH-A-PORT IDDD-related TEAE | 0 | 0 | 4 | 0
  IT administration process related TEAE | 4 | 3 | 1 | 1
  Severe TEAE | 2 | 3 | 1 | 1
  Serious TEAE | 5 | 4 | 3 | 2

2. Primary Outcome: Number of Participants With Clinical Laboratory Abnormalities Reported as Treatment Emergent Adverse Events (TEAEs)
Description: Clinical laboratory test included serum chemistry, hematology and urinalysis. Clinical laboratory abnormalities were recorded and reported as TEAE. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were defined as all AEs that occurred at or after the first dose of the investigational product or device implant surgery (whichever occurred earlier) and through the last follow-up date.
Time Frame: From start of study treatment up to Week 40
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Gamma-glutamyltransferase (GGT) increased | 2 | 1 | 1 | 0
  Alanine aminotransferase (ALT) increased | 1 | 1 | 0 | 1
  Aspartate aminotransferase (AST) increased | 0 | 1 | 1 | 0
  Blood iron decreased | 0 | 1 | 1 | 0
  Amylase increased | 0 | 1 | 1 | 0
  Blood alkaline phosphatase increased | 1 | 0 | 0 | 0
  Blood creatine phosphokinase increased | 0 | 0 | 0 | 3
  Hepatic enzymes increased | 0 | 0 | 0 | 1
  Eosinophil count increased | 0 | 1 | 1 | 0
  Eosinophilia | 0 | 2 | 0 | 0
  Mean cell volume decreased | 0 | 1 | 0 | 0
  Neutrophil count increased | 0 | 1 | 0 | 0
  White blood cell count increased | 0 | 1 | 0 | 0
  Lymphopenia | 0 | 1 | 0 | 0
  Leukocytosis | 0 | 1 | 0 | 0
  Proteinuria | 0 | 1 | 0 | 0

3. Primary Outcome: Number of Participants With Vital Sign Abnormalities Reported as Treatment Emergent Adverse Events (TEAEs)
Description: Vital sign assessments included blood pressure, heart rate, respiratory rate and body temperature. Vital sign abnormalities were recorded and reported as TEAE. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were defined as all AEs that occurred at or after the first dose of the investigational product or device implant surgery (whichever occurred earlier) and through the last follow-up date. Vital sign abnormalities included pyrexia which was considered as TEAE and was reported.
Time Frame: From start of study treatment up to Week 40
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 5 | 3 | 5 | 5

4. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities Reported as Treatment Emergent Adverse Events (TEAEs)
Description: 12-lead ECG was recorded and measured with the participant in rested supine position for at least 10 minutes. ECG abnormalities were recorded and reported as TEAE. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were defined as all AEs that occurred at or after the first dose of the investigational product or device implant surgery (whichever occurred earlier) and through the last follow-up date.
Time Frame: From start of study treatment up to Week 40
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Abnormalities in Physical Examination Reported as Treatment Emergent Adverse Events (TEAE)
Description: Complete physical examination included evaluation of the port and catheter track. Height or length and weight were recorded and used to calculate growth. Body weight and height measurements were used to calculate the body mass index (BMI). Head circumference was measured in uniform manner for all participants. Clinical significance was defined as any variation in physical findings that had medical relevance resulting in an alteration in medical care. Clinically significant abnormalities related to physical examination were recorded and reported as TEAE. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were defined as all AEs that occurred at or after the first dose of the investigational product or device implant surgery (whichever occurred earlier) and through the last follow-up date.
Time Frame: From start of study treatment up to Week 40
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants | 0 | 0 | 0 | 0

6. Primary Outcome: Number of Participants With Cerebrospinal Fluid (CSF) Chemistry Abnormalities Reported as Treatment Emergent Adverse Events (TEAEs)
Description: CSF chemistry assessments (including cell counts, glucose and protein) was measured. CSF chemistry abnormalities were recorded and reported as TEAE. An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. TEAEs were defined as all AEs that occurred at or after the first dose of the investigational product or device implant surgery (whichever occurred earlier) and through the last follow-up date.
Time Frame: From start of study treatment up to Week 40
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  CSF Protein Increased | 0 | 0 | 1 | 1
  CSF Albumin Increased | 0 | 0 | 1 | 0

7. Primary Outcome: Number of Participants With Positive Anti-SHP611 Antibodies in Cerebrospinal Fluid (CSF) and or Serum
Description: Number of participants with positive anti-SHP611 antibody results in serum and in CSF were reported. A participant was considered positive if they had at least 1 positive result during the study.
Time Frame: Baseline up to Week 40
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Serum anti-SHP611 antibody (Ab) positive | 4 | 3 | 1 | 2
  Serum neutralizing anti-SHP611 antibody positive | 3 | 2 | 1 | 1
  CSF anti-SHP611 antibody positive | 3 | 1 | 0 | 2
  CSF neutralizing anti-SHP611 antibody positive | 0 | 0 | 0 | 0
  Serum or CSF anti-SHP611 antibody positive | 4 | 3 | 1 | 2
  Serum and CSF anti-SHP611 antibody positive | 3 | 1 | 0 | 2
  Serum or CSF neutralizing anti-SHP611 Ab positive | 3 | 2 | 1 | 1
  Serum and CSF neutralizing anti-SHP611 Ab positive | 0 | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline in Motor Function Using Gross Motor Function Measure 88 (GMFM-88) Total Score at Week 40
Description: The GMFM-88 was used to measure motor function. The GMFM-88 item scores were used to calculate domain-specific percent score for each of the 5 GMFM-88 dimensions (lying and rolling; sitting; crawling and kneeling; standing; walking, running, and jumping), and a total GMFM-88 (percent) score was calculated based on each dimension score. Each of the 88 items was rated on a 4-point scale: 0=does not initiate; 1=initiates; 2=partially completes; and 3=completes. The GMFM-88 total scores ranged from 0% (no mobility) to a score of 100%, that is (i.e,) the score that can be obtained by an average 5-year-old or older child with normal motor abilities.
Time Frame: Baseline, Week 40
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: Score on a Scale
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Score on a Scale | -31.9 (8.76) | -29.0 (8.58) | -19.5 (8.54) | -18.1 (9.14)

9. Secondary Outcome: Number of Participants With Shift in Functional Endoscopic Evaluation of Swallowing (FEES) for Texture Utilized at Week 40
Description: The FEES assessment was performed to evaluate the structure and function of the upper throat during swallowing and for an assessment of aspiration risk. Each participant had this assessment performed at the clinical site using transnasal flexible laryngoscopy. FEES for texture utilized was evaluated. Data was presented only for the shifts observed.
Time Frame: Week 40
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Thin Liquids to Thin Liquids | 2 | 2 | 2 | 4
  Thin Liquids to Thickened Liquids | 1 | 2 | 0 | 0
  Thin Liquids to Puree Texture | 1 | 2 | 1 | 4
  Thin Liquids to Solids | 0 | 2 | 0 | 0
  Thickened Liquids to Thin Liquids | 1 | 2 | 1 | 1
  Thickened Liquids to Thickened Liquids | 0 | 2 | 3 | 0
  Thickened Liquids to Puree Texture | 1 | 2 | 3 | 1
  Thickened Liquids to Solids | 0 | 2 | 0 | 0
  Puree Texture to Thin Liquids | 1 | 2 | 3 | 2
  Puree Texture to Thickened Liquids | 1 | 2 | 2 | 0
  Puree Texture to Puree Texture | 3 | 4 | 4 | 3
  Puree Texture to Solids | 0 | 2 | 0 | 0
  Solids to Thin Liquids | 0 | 2 | 0 | 1
  Solids to Thickened Liquids | 0 | 2 | 0 | 0
  Solids to Puree Texture | 0 | 2 | 0 | 1
  Solids to Solids | 0 | 2 | 0 | 0

10. Secondary Outcome: Number of Participants With Shift in Functional Endoscopic Evaluation of Swallowing for Feeding Assessment (Laryngeal Penetration) at Week 40
Description: The FEES assessment was performed to evaluate the structure and function of the upper throat during swallowing and for an assessment of aspiration risk. Each participant had this assessment performed at the clinical site using transnasal flexible laryngoscopy. Feeding assessment for laryngeal penetration was assessed. Data was presented only for the shifts observed. Here TL refers to thin liquids, THL refers to thickened liquids, PT refers to puree texture, WCC refers to with cough and clearance and WCNC refers to with cough and no clearance.
Time Frame: Week 40
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Normal to Normal (TL) | 0 | 0 | 2 | 1
  Normal to Without Cough (TL) | 0 | 0 | 0 | 1
  Without Cough to Without Cough (TL) | 1 | 0 | 0 | 0
  WCC to Without Cough (TL) | 1 | 0 | 0 | 0
  WCC to WCC (TL) | 0 | 2 | 0 | 1
  Normal to WCC (THL) | 0 | 0 | 1 | 0
  Without Cough to Normal (THL) | 0 | 0 | 1 | 0
  WCC to Normal (THL) | 0 | 0 | 1 | 0
  WCC to WCC (THL) | 0 | 2 | 0 | 0
  Normal to Normal (PT) | 0 | 1 | 1 | 1
  Normal to WCC (PT) | 0 | 0 | 1 | 0
  Normal to WCNC (PT) | 1 | 0 | 0 | 0
  Without Cough to Normal (PT) | 0 | 0 | 2 | 0
  Without Cough to WCC (PT) | 1 | 0 | 0 | 0
  WCC to Normal (PT) | 0 | 0 | 0 | 1
  WCC to WCC (PT) | 0 | 2 | 0 | 0
  WCNC to Normal (PT) | 0 | 1 | 0 | 0
  WCNC to Without Cough (PT) | 1 | 0 | 0 | 0
  WCC to WCC (Solids) | NA — Data was not available for this texture as the assessment was considered normal. | 2 | NA — Data was not available for this texture as the assessment was considered normal. | NA — Data was not available for this texture as the assessment was considered normal.

11. Secondary Outcome: Number of Participants With Shift in Functional Endoscopic Evaluation of Swallowing for Feeding Assessment (Aspiration Through Vocal Cords) at Week 40
Description: The FEES assessment was performed to evaluate the structure and function of the upper throat during swallowing and for an assessment of aspiration risk. Each participant had this assessment performed at the clinical site using transnasal flexible laryngoscopy. Feeding assessment for aspiration through vocal cords were assessed. Data was presented only for the shifts observed. Here TL refers to thin liquids, THL refers to thickened liquids, PT refers to puree texture, WCC refers to with cough and clearance and WCNC refers to with cough and no clearance.
Time Frame: Week 40
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Normal to Normal (TL) | 0 | 0 | 2 | 3
  Without Cough to Without Cough (TL) | 1 | 0 | 0 | 0
  WCC to WCC (TL) | 0 | 2 | 0 | 0
  Normal to Normal (THL) | 0 | 0 | 1 | 0
  Without Cough to Normal (THL) | 0 | 0 | 1 | 0
  WCC to Normal (THL) | 0 | 0 | 1 | 0
  WCC to WCC (THL) | 0 | 2 | 0 | 0
  Normal to Normal (PT) | 0 | 2 | 2 | 2
  Without Cough to Normal (PT) | 0 | 0 | 2 | 0
  WCC to WCC (PT) | 0 | 2 | 0 | 0
  WCNC to Normal (PT) | 1 | 0 | 0 | 0
  WCC to WCC (Solids) | NA — Data was not available for this texture as the assessment was considered normal. | 2 | NA — Data was not available for this texture as the assessment was considered normal. | NA — Data was not available for this texture as the assessment was considered normal.

12. Secondary Outcome: Number of Participants With Shift in Functional Endoscopic Evaluation of Swallowing for Dose Residue Clear After Subsequent Swallowing at Week 40
Description: The FEES assessment was performed to evaluate the structure and function of the upper throat during swallowing and for an assessment of aspiration risk. Each participant had this assessment performed at the clinical site using transnasal flexible laryngoscopy. FEES for dose residue clear after subsequent swallowing was assessed. Data was presented only for the shifts observed. Here TL refers to thin liquids, THL refers to thickened liquids, PT refers to puree texture.
Time Frame: Week 40
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Normal to Normal (TL) | 0 | 0 | 1 | 0
  Normal to Yes (TL) | 0 | 0 | 1 | 0
  Yes to Yes (TL) | 1 | 2 | 0 | 1
  Yes to No (TL) | 0 | 0 | 0 | 1
  No to Yes (TL) | 0 | 0 | 0 | 1
  No to No (TL) | 1 | 0 | 0 | 0
  Normal to Yes (THL) | 0 | 0 | 2 | 0
  Yes to Normal (THL) | 0 | 0 | 1 | 0
  Yes to Yes (THL) | 0 | 2 | 0 | 0
  Normal to Normal (PT) | 0 | 1 | 0 | 1
  Normal to Yes (PT) | 0 | 0 | 2 | 0
  Normal to No (PT) | 1 | 0 | 0 | 0
  Yes to Normal (PT) | 0 | 0 | 1 | 0
  Yes to Yes (PT) | 1 | 2 | 0 | 1
  Yes to No (PT) | 1 | 0 | 0 | 0
  No to Normal (PT) | 0 | 1 | 1 | 0
  Yes to Yes (Solids) | NA — Data was not available for this texture as the assessment was considered normal. | 2 | NA — Data was not available for this texture as the assessment was considered normal. | NA — Data was not available for this texture as the assessment was considered normal.

13. Secondary Outcome: Number of Participants With Shift in Functional Endoscopic Evaluation of Swallowing for Aspiration Risk at Week 40
Description: The FEES assessment was performed to evaluate the structure and function of the upper throat during swallowing and for an assessment of aspiration risk. Each participant had this assessment performed at the clinical site using transnasal flexible laryngoscopy. FEES for aspiration risk was assessed. Data was presented only for the shifts observed. Here TL refers to thin liquids, THL refers to thickened liquids, PT refers to puree texture, WCC refers to with cough and clearance and WCNC refers to with cough and no clearance.
Time Frame: Week 40
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Low to Low (TL) | 2 | 2 | 2 | 3
  Low to High (TL) | 0 | 0 | 0 | 1
  Low to Low (THL) | 0 | 2 | 3 | 0
  Low to Low (PT) | 1 | 3 | 3 | 3
  Low to High (PT) | 1 | 0 | 0 | 0
  Moderate to Low (PT) | 0 | 1 | 1 | 0
  Moderate to Moderate (PT) | 1 | 0 | 0 | 0
  Low to Low (Solids) | NA — Data was not available for this texture as the assessment was considered normal. | 2 | NA — Data was not available for this texture as the assessment was considered normal. | NA — Data was not available for this texture as the assessment was considered normal.

14. Secondary Outcome: Number of Participants With Change in Nerve Conduction as Measured by Electroneurography (ENG) Assessments by Categorized Amplitude Values at Week 40
Description: Evaluation of peripheral nerve function by ENG studies was performed to measure nerve conduction velocity (NCV), amplitude (AMP),distal latency (DL), and F-wave latency. Categorized amplitude values were assessed. Data was presented only for number of participants who reported change in amplitude greater than (>) 0.
Time Frame: Baseline, Week 40
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  Median Motor Wrist Amplitude (Baseline) | 6 | 5 | 5 | 6
  Median Motor Wrist Amplitude (Week 40) | 3 | 5 | 6 | 5
  Median Motor Elbow Amplitude (Baseline) | 0 | 2 | 4 | 6
  Median Motor Elbow Amplitude (Week 40) | 0 | 4 | 6 | 4
  Median Sensory Wrist Amplitude (Baseline) | 2 | 3 | 4 | 4
  Median Sensory Wrist Amplitude (Week 40) | 1 | 5 | 3 | 3
  Peroneal Motor Fibular Head Amplitude (Baseline) | 0 | 2 | 4 | 6
  Peroneal Motor Fibular Head Amplitude (Week 40) | 0 | 4 | 5 | 4
  Peroneal Motor Ankle Amplitude (Baseline) | 6 | 5 | 5 | 6
  Peroneal Motor Ankle Amplitude (Week 40) | 4 | 5 | 5 | 4
  Sural Sensory B-point (Baseline) | 2 | 2 | 3 | 4
  Sural Sensory B-point (Week 40) | 2 | 2 | 3 | 4
  Tibial Motor Ankle Amplitude (Baseline) | 4 | 3 | 3 | 3
  Tibial Motor Ankle Amplitude (Week 40) | 2 | 3 | 4 | 1
  Tibial Motor Knee Amplitude (Baseline) | 0 | 0 | 3 | 3
  Tibial Motor Knee Amplitude (Week 40) | 0 | 2 | 4 | 1
  Ulnar Motor Wrist Amplitude (Baseline) | 4 | 3 | 3 | 3
  Ulnar Motor Wrist Amplitude (Week 40) | 2 | 3 | 3 | 1
  Ulnar Motor Elbow Amplitude (Baseline) | 0 | 0 | 3 | 3
  Ulnar Motor Elbow Amplitude (Week 40) | 0 | 2 | 3 | 1

15. Secondary Outcome: Number of Participants With Change in Nerve Conduction as Measured by Electroneurography (ENG) Assessments by Categorized Nerve Conduction Velocity at Week 40
Description: Evaluation of peripheral nerve function by ENG studies was performed to measure nerve conduction velocity (NCV), amplitude (AMP),distal latency (DL), and F-wave latency. Categorized nerve conduction velocity values were assessed. Data was presented only for number of participants who reported change in nerve conduction velocity > 0. Here MME refers to median motor elbow, WCV for wrist conduction velocity, PMA for peroneal motor ankle, FHCV to fibular head conduction velocity, TMA for tibial motor ankle, KCV for knee conduction velocity and UME for ulnar motor elbow,
Time Frame: Baseline, Week 40
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  MME to WCV (Baseline) | 6 | 6 | 6 | 6
  MME to WCV (Week 40) | 3 | 5 | 6 | 5
  PMA to FHCV (Baseline) | 6 | 6 | 6 | 6
  PMA to FHCV (Week 40) | 4 | 5 | 5 | 4
  TMA to KCV (Baseline) | 4 | 4 | 4 | 3
  TMA to KCV (Week 40) | 2 | 3 | 4 | 1
  UME to WCV (Baseline) | 4 | 4 | 4 | 3
  UME to WCV (Week 40) | 2 | 3 | 3 | 1

16. Secondary Outcome: Number of Participants With Change in Nerve Conduction as Measured by Electroneurography (ENG) Assessments by Categorized Distal Latency at Week 40
Description: Evaluation of peripheral nerve function by ENG studies was performed to measure nerve conduction velocity (NCV), amplitude (AMP),distal latency (DL), and F-wave latency. Categorized amplitude values were assessed. Data was presented only for number of participants who reported change in distal latency > 0. Here MMW refers to median motor wrist, APB for abductor pollicis brevis, MSW for median sensory wrist, DDL for digit distal latency, PMA for peroneal motor ankle, EDB for extensor digitorum brevis, SSB-point DL for sural sensory B-point distal latency, TMA for tibial motor ankle, abductor hallucis for AH distal latency and, UMW for ulnar motor wrist.
Time Frame: Baseline, Week 40
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Participants
  MMW to APB distal latency (Baseline) | 6 | 5 | 5 | 6
  MMW to APB distal latency (Week 40) | 3 | 5 | 6 | 5
  MSW to DDL (Baseline) | 0 | 1 | 2 | 3
  MSW to DDL (Week 40) | 0 | 3 | 2 | 3
  PMA to EDB Distal Latency (Baseline) | 6 | 5 | 5 | 6
  PMA to EDB Distal Latency (Week 40) | 4 | 5 | 5 | 3
  SS B-Point Distal Latency (Baseline) | 2 | 2 | 2 | 3
  SS B-Point Distal Latency (Week 40) | 1 | 2 | 1 | 4
  TMA to AH Distal Latency (Baseline) | 0 | 0 | 3 | 3
  TMA to AH Distal Latency (Week 40) | 0 | 2 | 4 | 0
  UMW to ADM Distal Latency (Baseline) | 4 | 3 | 3 | 3
  UMW to ADM Distal Latency (Week 40) | 2 | 3 | 3 | 1

17. Secondary Outcome: Change From Baseline in Adaptive Behavior Composite Standard Score as Measured by Vineland Adaptive Behavior Scales, Second Edition (VABS-II) at Week 40
Description: The VABS-II test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. This test measures the following 4 key domains: communication, daily living skills, socialization, motor skills, and the adaptive behavior composite (ABC) (a composite of the other 4 domain). Items in each domain are rated as either 0 (does not), 1(sometimes) or 2(independently) performs a given behavior or skill. The 4 domain standard scores range from 20-160 and higher scores indicate a higher level of functioning. ABC scores have a mean of 100 and a standard deviation of 15 (range = 20 to 160) and higher scores indicate a higher level of functioning. A positive change value indicates improvement in adaptive functioning.
Time Frame: Baseline, Week 40
Population: Safety set consisted of participants who received at least 1 dose of investigational product or underwent device implant surgery. Participants from SHP611 10 mg and SHP611 30 mg were excluded from the analysis. Since, analysis was planned for participants received SHP611 100 mg with different manufacturing processes (Process A and B).
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6
Score on a scale
  Communication(Baseline): number analyzed (Participants) | 1 | 3
  Communication(Baseline) | 52.0 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 97.3 (2.52)
  Communication(Week 40): number analyzed (Participants) | 1 | 3
  Communication(Week 40) | -10.0 (NA) — Standard deviation was not calculated due to insufficient number of participants. | -25.0 (18.19)
  Daily Living Skills(Baseline): number analyzed (Participants) | 2 | 3
  Daily Living Skills(Baseline) | 49.0 (1.41) | 80.3 (9.02)
  Daily Living Skills(Week 40): number analyzed (Participants) | 2 | 3
  Daily Living Skills(Week 40) | -4.0 (5.66) | -27.0 (19.47)
  Socialization(Baseline): number analyzed (Participants) | 2 | 3
  Socialization(Baseline) | 50.0 (1.41) | 86.0 (3.61)
  Socialization(Week 40): number analyzed (Participants) | 2 | 3
  Socialization(Week 40) | -0.5 (0.71) | -18.0 (17.09)
  Motor Skills(Baseline): number analyzed (Participants) | 2 | 3
  Motor Skills(Baseline) | 31.0 (0.00) | 83.7 (24.83)
  Motor Skills(Week 40): number analyzed (Participants) | 2 | 3
  Motor Skills(Week 40) | 6.0 (16.97) | -43.3 (23.18)
  Adaptive Behavior CSS(Baseline): number analyzed (Participants) | 1 | 3
  Adaptive Behavior CSS(Baseline) | 43.0 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 84.0 (10.54)
  Adaptive Behavior CSS(Week 40): number analyzed (Participants) | 1 | 3
  Adaptive Behavior CSS(Week 40) | -5.0 (NA) — Standard deviation was not calculated due to insufficient number of participants. | -25.3 (16.44)

18. Secondary Outcome: Change From Baseline in Domain-specific Caregiver Observed Metachromatic Leukodystrophy (MLD) Functioning and Outcomes Reporting Tool (COMFORT) Scores at Week 40
Description: COMFORT questionnaire was used to assess health status and the impact of disease on the ability of participants with MLD to carry out activities of daily life. The questionnaire was organized by 8 domains (ie, personal care; positioning, transfer, or mobility; eating; pain and discomfort during the day; sleep; emotions; communication; and play and leisure activities). The COMFORT scores range from 0 to 100, with higher scores indicating a decline in the functioning.
Time Frame: Baseline, Week 40
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6
Score on a scale
  Communication (Baseline): number analyzed (Participants) | 5 | 6
  Communication (Baseline) | 27.3 (13.27) | 16.9 (8.65)
  Communication (Week 40): number analyzed (Participants) | 5 | 6
  Communication (Week 40) | 24.7 (26.81) | 21.4 (20.92)
  Eating difficulty (Baseline): number analyzed (Participants) | 5 | 6
  Eating difficulty (Baseline) | 21.1 (22.94) | 2.4 (5.77)
  Eating difficulty (Week 40): number analyzed (Participants) | 5 | 6
  Eating difficulty (Week 40) | 25.1 (22.44) | 11.8 (10.29)
  Emotions (Baseline): number analyzed (Participants) | 5 | 6
  Emotions (Baseline) | 60.0 (9.13) | 55.6 (12.55)
  Emotions (Week 40): number analyzed (Participants) | 5 | 6
  Emotions (Week 40) | -15.0 (21.57) | -1.4 (6.27)
  Pain and discomfort during the day (Baseline): number analyzed (Participants) | 5 | 6
  Pain and discomfort during the day (Baseline) | 16.6 (10.16) | 6.9 (11.05)
  Pain and discomfort during the day (Week 40): number analyzed (Participants) | 5 | 6
  Pain and discomfort during the day (Week 40) | 13.5 (15.23) | 0.0 (11.74)
  Personal care (Baseline): number analyzed (Participants) | 5 | 6
  Personal care (Baseline) | 48.0 (21.26) | 36.0 (17.99)
  Personal care (Week 40): number analyzed (Participants) | 5 | 6
  Personal care (Week 40) | 18.1 (37.94) | 7.3 (18.95)
  Play and leisure activities (Baseline): number analyzed (Participants) | 5 | 6
  Play and leisure activities (Baseline) | 46.0 (19.81) | 16.7 (16.33)
  Play and leisure activities (Week 40): number analyzed (Participants) | 5 | 6
  Play and leisure activities (Week 40) | 1.0 (28.15) | 30.0 (25.88)
  Positioning, transfer or mobility (Baseline): number analyzed (Participants) | 5 | 6
  Positioning, transfer or mobility (Baseline) | 42.2 (19.44) | 18.0 (18.80)
  Positioning, transfer or mobility (Week 40): number analyzed (Participants) | 5 | 6
  Positioning, transfer or mobility (Week 40) | 6.7 (21.82) | 8.8 (13.14)
  Sleep (Baseline): number analyzed (Participants) | 5 | 6
  Sleep (Baseline) | 11.9 (5.52) | 18.9 (6.52)
  Sleep (Week 40): number analyzed (Participants) | 5 | 6
  Sleep (Week 40) | 6.8 (17.08) | 4.5 (15.60)

19. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of SHP611
Description: Cmax is the maximum observed serum concentration of SHP611.
Time Frame: Baseline: Predose, 0.5, 1, 2, 4, 8, 12, 24, 48 hours postdose; Week 38: Predose, 0.5, 1, 2, 4, 8, 12, 24, 48 hours postdose
Population: Pharmacokinetic (PK) set consisted of participants who received at least 1 dose of investigational product and had at least 1 measurable serum concentration or 1 measurable CSF concentration of SHP611.
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Nanogram per milliliter (ng/mL)
  Baseline: number analyzed (Participants) | 6 | 6 | 6 | 5
  Baseline | 214.53 (162.104) | 500.83 (260.978) | 715.17 (339.856) | 799.60 (494.452)
  Week 38: number analyzed (Participants) | 2 | 5 | 4 | 4
  Week 38 | 157.50 (36.062) | 275.40 (156.329) | 888.75 (225.457) | 1494.83 (1297.295)

20. Secondary Outcome: Time to Reach Maximum Observed Drug Concentration (Tmax) of SHP611 in Plasma
Description: Tmax is the time to reach maximum observed drug concentration of SHP611 during a dosing interval.
Time Frame: as for outcome 19
Population: PK set consisted of participants who received at least 1 dose of investigational product and had at least 1 measurable serum concentration or 1 measurable CSF concentration of SHP611.
Measure: Mean (Standard Deviation); unit: Hour (h)
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Hour (h)
  Baseline: number analyzed (Participants) | 6 | 6 | 6 | 5
  Baseline | 7.06 (1.086) | 6.81 (3.462) | 5.97 (4.802) | 9.61 (8.344)
  Week 38: number analyzed (Participants) | 2 | 5 | 4 | 4
  Week 38 | 5.08 (1.450) | 11.22 (1.780) | 18.16 (11.661) | 7.02 (3.824)

21. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of SHP611
Description: The AUC0-inf is the area under the concentration-time curve from time zero to infinity of SHP611.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Hour * nanogram/milliliter (h*ng/mL)
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Hour * nanogram/milliliter (h*ng/mL)
  Baseline: number analyzed (Participants) | 1 | 4 | 2 | 3
  Baseline | 4355 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 10105 (3307.4) | 22123 (4217.4) | 23117 (10380.1)
  Week 38: number analyzed (Participants) | 1 | 1 | 0 | 2
  Week 38 | 2767 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 9589 (NA) — Standard deviation was not calculated due to insufficient number of participants. |  | 48648 (6906.8)

22. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to the Time of the Last Quantifiable Concentration (AUC0-last) of SHP611
Description: AUC0-last is the area under the concentration-time curve from the time of dosing to the last measurable concentration of SHP611.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: hour * nanogram per milliliter (h*ng/mL)
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour * nanogram per milliliter (h*ng/mL)
  Baseline: number analyzed (Participants) | 6 | 6 | 6 | 5
  Baseline | 2532 (1178.4) | 8738 (3106.4) | 15022 (10755.2) | 16288 (10691.4)
  Week 38: number analyzed (Participants) | 2 | 5 | 4 | 4
  Week 38 | 1972 (211.5) | 6156 (3904.5) | 24820 (16954.3) | 29219 (21261.5)

23. Secondary Outcome: Area Under the Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24) of SHP611
Description: Area under the concentration-time curve over the interval from 0 to 24 hours after dosing of SHP611.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: hour * nanogram per milliliter (h*ng/mL)
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
hour * nanogram per milliliter (h*ng/mL)
  Baseline: number analyzed (Participants) | 6 | 6 | 5 | 5
  Baseline | 2530 (1178.0) | 6258 (2995.3) | 11918 (6376.1) | 13114 (8012.0)
  Week 38: number analyzed (Participants) | 2 | 4 | 3 | 3
  Week 38 | 1960 (224.0) | 4596 (2316.1) | 18264 (2162.7) | 31115 (15805.6)

24. Secondary Outcome: First Order Rate Constant (Lambda z) Associated With the Terminal (Log-linear) Portion of the Curve for SHP611
Description: Lambda z is first order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Per hour (/h)
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Per hour (/h)
  Baseline: number analyzed (Participants) | 1 | 4 | 2 | 3
  Baseline | 0.0934 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 0.0561 (0.01900) | 0.0461 (0.02439) | 0.0607 (0.01949)
  Week 38: number analyzed (Participants) | 1 | 1 | 0 | 2
  Week 38 | 0.0506 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 0.0640 (NA) — Standard deviation was not calculated due to insufficient number of participants. |  | 0.0857 (0.04415)

25. Secondary Outcome: Terminal Elimination Half Life (t1/2) of SHP611
Description: The t1/2 is the time in hours required for the concentration of the drug to reach half of its original value.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Hour (h)
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Hour (h)
  Baseline: number analyzed (Participants) | 1 | 4 | 2 | 3
  Baseline | 7.42 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 13.60 (4.932) | 17.47 (9.238) | 12.34 (4.373)
  Week 38: number analyzed (Participants) | 1 | 1 | 0 | 2
  Week 38 | 13.70 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 10.83 (NA) — Standard deviation was not calculated due to insufficient number of participants. |  | 9.32 (4.800)

26. Secondary Outcome: Total Body Clearance (CL/F) After Intrathecal Administration of SHP611
Description: CL/F was defined as the total body clearance of the drug for extravascular administration divided by the fraction of dose absorbed.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Liter per hour (L/h)
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Liter per hour (L/h)
  Baseline: number analyzed (Participants) | 1 | 4 | 2 | 3
  Baseline | 2.30 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 3.25 (1.185) | 4.60 (0.878) | 5.28 (3.179)
  Week 38: number analyzed (Participants) | 1 | 1 | 0 | 2
  Week 38 | 3.61 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 3.13 (NA) — Standard deviation was not calculated due to insufficient number of participants. |  | 2.08 (0.295)

27. Secondary Outcome: Volume of Distribution (Vz/F) After Intrathecal Administration of SHP611
Description: Volume of distribution was associated with the terminal slope following extravascular administration of SHP611 divided by the fraction of dose absorbed.
Time Frame: as for outcome 19
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Liter (L)
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Liter (L)
  Baseline: number analyzed (Participants) | 1 | 4 | 2 | 3
  Baseline | 24.58 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 69.97 (49.912) | 121.88 (83.481) | 106.95 (100.026)
  Week 38: number analyzed (Participants) | 1 | 1 | 0 | 2
  Week 38 | 71.41 (NA) — Standard deviation was not calculated due to insufficient number of participants. | 48.88 (NA) — Standard deviation was not calculated due to insufficient number of participants. |  | 28.95 (18.345)

28. Secondary Outcome: Concentration of SHP611 in Cerebrospinal Fluid
Description: Concentration of SHP611 in CSF was determined using validated enzyme-linked immunosorbent assay (ELISA) method.
Time Frame: Baseline, 4, 8, 12, 16, 20, 24, 28, 32, 36, and 40 weeks
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Nanogram per milliliter (ng/mL)
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
Number analyzed (Participants) | 6 | 6 | 6 | 6
Nanogram per milliliter (ng/mL)
  Baseline: number analyzed (Participants) | 6 | 6 | 6 | 5
  Baseline | 280.00 (685.857) | 0 (0) | 0 (0) | 0 (0)
  Week 4: number analyzed (Participants) | 6 | 6 | 6 | 4
  Week 4 | 182.93 (165.913) | 78.00 (102.516) | 2935.17 (2632.398) | 6152.50 (6546.986)
  Week 8: number analyzed (Participants) | 6 | 6 | 5 | 4
  Week 8 | 85.47 (79.316) | 1854.07 (2633.858) | 4171.20 (4874.122) | 3825.00 (2182.056)
  Week 12: number analyzed (Participants) | 5 | 6 | 6 | 5
  Week 12 | 57.50 (57.365) | 1556.17 (1557.666) | 2310.00 (2544.814) | 2304.00 (2155.558)
  Week 16: number analyzed (Participants) | 6 | 6 | 6 | 5
  Week 16 | 93.83 (147.188) | 2805.68 (3499.878) | 2395.00 (1550.648) | 2606.20 (1212.857)
  Week 20: number analyzed (Participants) | 6 | 6 | 6 | 3
  Week 20 | 112.78 (143.216) | 1364.65 (2784.474) | 5182.50 (5081.080) | 4423.33 (4195.406)
  Week 24: number analyzed (Participants) | 6 | 6 | 6 | 5
  Week 24 | 132.57 (235.783) | 802.67 (903.025) | 5402.50 (7352.246) | 7914.60 (8243.114)
  Week 28: number analyzed (Participants) | 5 | 6 | 6 | 4
  Week 28 | 525.06 (874.710) | 3274.62 (4493.212) | 6273.83 (6839.101) | 3682.58 (4331.130)
  Week 32: number analyzed (Participants) | 5 | 6 | 5 | 5
  Week 32 | 70.12 (126.513) | 573.62 (376.224) | 1831.40 (988.294) | 6110.00 (4099.500)
  Week 36: number analyzed (Participants) | 5 | 6 | 6 | 3
  Week 36 | 72.40 (125.574) | 1046.05 (1087.321) | 3917.50 (4650.791) | 3116.67 (336.502)
  Week 40: number analyzed (Participants) | 6 | 2 | 6 | 4
  Week 40 | 659.15 (1602.414) | 243.60 (313.107) | 2931.83 (4098.389) | 6663.75 (7947.148)

ADVERSE EVENTS:
Time Frame: From start of study treatment up to safety follow up (Week 42)
Groups:
- SHP611 10 mg (Process A): Participants received 10 mg dose of SHP611 (HGT-1110, rhASA) EOW by IDDD for 38 weeks.
- SHP611 30 mg (Process A): Participants received 30 mg dose of SHP611 (HGT-1110, rhASA) EOW by IDDD for 38 weeks.
- SHP611 100 mg (Process A); SHP611 100 mg (Process B): Participants received 100 mg dose of SHP611 (HGT-1110, rhASA) EOW by IDDD for 38 weeks.
Arm/Group | SHP611 10 mg (Process A) | SHP611 30 mg (Process A) | SHP611 100 mg (Process A) | SHP611 100 mg (Process B)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 5/6 | 4/6 | 3/6 | 2/6
Other Adverse Events (participants affected / at risk) | 6/6 | 6/6 | 6/6 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP611 10 mg (Process A) (N=6) | SHP611 30 mg (Process A) (N=6) | SHP611 100 mg (Process A) (N=6) | SHP611 100 mg (Process B) (N=6)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Device failure (General disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Device malfunction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Implant site effusion (General disorders) | 1 (1) | 0 (0) | 1 (3) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gamma-Glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 1 (3) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Muscle spasticity (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SHP611 10 mg (Process A) (N=6) | SHP611 30 mg (Process A) (N=6) | SHP611 100 mg (Process A) (N=6) | SHP611 100 mg (Process B) (N=6)
Eosinophilia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Kyphosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lordosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Tendinous contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendon disorder (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual acuity reduced (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 4 (7) | 3 (3) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (2) | 1 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Gingivitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (4) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary duct obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 4 (5) | 5 (7) | 4 (11) | 2 (6)
Asthenia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Complication of device removal (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Crying (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device dislocation (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Device malfunction (General disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gait disturbance (General disorders) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Implant site cyst (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Implant site effusion (General disorders) | 1 (1) | 0 (0) | 3 (6) | 1 (1)
Implant site pain (General disorders) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 5 (15) | 3 (17) | 5 (6) | 5 (11)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Talipes (Congenital, familial and genetic disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (6) | 1 (1) | 1 (1) | 1 (2)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 2 (3) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rhinitis (Infections and infestations) | 2 (3) | 2 (3) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 3 (5) | 1 (1) | 2 (5)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (2) | 0 (0) | 2 (3) | 0 (0)
Viral pharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endotracheal intubation complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Incision site oedema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural oedema (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 2 (2) | 3 (3) | 5 (5)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrong technique in drug usage process (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Albumin csf increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amylase increased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Blood iron decreased (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Blood pressure increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Csf lymphocyte count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Csf mononuclear cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Csf protein increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Csf white blood cell count increased (Investigations) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Eosinophil count increased (Investigations) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
Gamma-Glutamyltransferase increased (Investigations) | 2 (4) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Mean cell volume decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Red blood cells csf positive (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cytolytic hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iron deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Areflexia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebellar syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Clonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Disturbance in attention (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dystonia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Hypotonia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Motor dysfunction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasticity (Nervous system disorders) | 4 (4) | 2 (3) | 1 (1) | 2 (2)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 2 (3) | 3 (3) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Speech disorder developmental (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abnormal behaviour (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased eye contact (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Initial insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 3 (3) | 1 (1) | 0 (0) | 2 (3)
Balanitis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hirsutism (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Keloid scar (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (3) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2015-08-25): https://cdn.clinicaltrials.gov/large-docs/28/NCT01510028/Prot_001.pdf
  • Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/28/NCT01510028/SAP_000.pdf